Queen Square MS Centre - UCL Institute of Neurology



Investigator: Professor Richard Nicholas

**Centre Number:** 

**Contact for Queries:** 

If you have any questions about this study, you can contact:

Daytime: 02031081955

Out of hours (emergency): 07970479797

The National Hospital for Neurology & Neurosurgery Queen Square London WC1N 3BG

## **Consent Form for the Simvastatin in PMS Study (MS-OPT)**

Sponsor Reference number: 16/0730

Version 1.3 dated 08/09/20

Study title: A double-blind, randomised, placebo-controlled single site study of high dose simvastatin treatment for progressive multiple sclerosis: impact on vascular perfusion and oxidative damage.

| Name of Researcher (PI): | |
|--------------------------|---------|
| Sponsor Study Number: | 16/0730 |
| Site: | |
| Participant Number: | |

Please initial each box

| 1. | I have read and understood the patient information leaflet (version 1.4 dated 08 Sept 2020) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. |
|---|---|
| 2. | I understand that my participation in this study is voluntary and that I am free to withdraw from the study at any time, without giving any reason, without my medical care or legal rights being affected. |
| 3. | As described in the study information leaflet, I understand that sections of my medical notes may be looked at by responsible individuals from CCTU, institutions acting on their behalf or regulatory authorities where it is relevant to my taking part in research. I give permission for these individuals to have access to my records. |
| 4. | As described in the study information leaflet, I understand that <b>non identifiable</b> data collected in the study may be sent to third parties (e.g. pharmaceutical companies or other academic institutions) for research, safety monitoring or licensing purposes and that this may involve some data being transferred within the European Union. |
| 5. | |

| | 6. As described in the study information leaflet, I agree to my GP and/or consultant being informed about my participation in the study. | | |
|---|---|---|---|
| 7. | sample stored for the purpose of future research for up to 10 years from the date of my consent. | | |
| 8. | | | |
| 9. | I freely agree to take part in thi | is study. | |
| Ple | ease print and sign your name | e below and add today's date: | |
| Na | me of patient | Signature | Date |
| | me of patient me of person taking consent | Signature | Date |
| <br>Na | ·<br> | Signature | |
| Na<br>N.I | me of person taking consent 3. The patient must date his/her | Signature | Date |